CLINICAL TRIAL: NCT01741909
Title: Can the Cost of Azythromycin in be Reduced in Hospitalized Patients With Community Acquired Pneumonia by Quick Transfer From Intravenous to Oral Therapy?
Brief Title: Reducing Cost of Azythromycin by Transferring From IV to Oral Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to recruiting issues
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Lee Goldstein, Lee Goldstein MD, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMC-85-12-CTIL
Record Dates: First submitted 2012-12-02; First posted 2012-12-05 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Pneumonia
Keywords: azythromycin; community acquired pneumonia; intravenous; oral
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Before, After (Experimental): The intervention is educational
  Interventions: Behavioral: education

INTERVENTIONS:
Behavioral: education — after a baseline period, shorter intravenous treatment will be promoted by mail, posters, lectures, and pharmacy monitoring of treatment

SUMMARY:
Intravenous Azythromycin therapy is considerably more expensive than oral therapy. The investigators believe that intravenous therapy is prolonged more that necessary and that oral therapy can be used much earlier in the course of the disease. The investigators plan to check if that statement is true and intervene in order to shorten the intravenous therapy.

DETAILED DESCRIPTION:
The study will be performed in two stages. First a retrospective review of medical files of 50 patients hospitalized in the Haemek Medical Center with severe community acquired pneumonia, treated with azythromycin. The files will be reviewed for the criteria clinical improvement, and for azythromycin therapy, oral or intravenous.

The results of this review will help us define the appropriate behavioral intervention in order to cause doctors to transfer from IV to PO therapy at the earliest appropriate time. An intervention such as posters, pharmacy overseeing etc will be introduced. 3 months after the intervention, an additional 50 files of pneumonia patients treated with azythromycin will be reviewed in order to check the efficacy of the intervention.

The Review board and the NIH will be updated about the intervention, as soon as the investigators have decided what intervention is appropriate

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized with community acquired pneumonia treated by azythromycin

Exclusion Criteria:

* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
length of intravenous azythromycin treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lee H Goldstein, MD, Principal Investigator — haemek medical center
Locations (1):
- Haemek Medical Center, Afula, Israel